CLINICAL TRIAL: NCT03384888
Title: Neurostimulation Applied to Fibromyalgia
Acronym: NeuroFibro
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Géssika Araújo de Melo, Eliane Araújo de Oliveira, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Eliane Araújo de Oliveira
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia, Neurostimulation, TDCS
MeSH Terms: conditions — Fibromyalgia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The parallel clinical trial simultaneously compares two groups of individuals, one of which receives the intervention of interest and the other is a control group (sham).
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ano-M1-cat-SO5 tDCS (Experimental): Participants will receive active transcranial direct current stimulation (tDCS) (active tDCS). The electrodes will be placed on left M1 for anodic stimulation and on the right supraorbital region for cathodic stimulation on 5 consecutive days.
  Interventions: Device: Active tDCS
- ano-M1-cat-SO10 tDCS (Experimental): Participants will receive active transcranial direct current stimulation (active tDCS). The electrodes will be placed on left M1 for anodic stimulation and on the right supraorbital region for cathodic stimulation on 10 consecutive days.
  Interventions: Device: Active tDCS
- Sham tDCS (Sham Comparator): Participants who receive stimulation of the simulated type (sham tDCS), following the protocol of the ano-M1-cat-SO5 group.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — Transcranial direct current stimulation Duration: 20 minutes; Intensity: 2 mA (miliamps); Placement of the electrodes: anode over the left M1 and cathode region over the right supraorbital region.
  Other Names: Transcranial direct current stimulation
  Arms: ano-M1-cat-SO10 tDCS; ano-M1-cat-SO5 tDCS
Device: Sham tDCS — Sham Transcranial direct current stimulation The procedure is the same as for active tDCS, but the stimulation is non-active / sham.
  Other Names: Transcranial direct current stimulation
  Arms: Sham tDCS

SUMMARY:
NeuroFibro is a double-blind, randomized, placebo-controlled clinical trial, using neurostimulation in women with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* (1) diagnosis of fibromyalgia, according to the American College of Rheumatology criteria;
* (2) been diagnosed for at least three months;
* (3) be female;
* (4) be in the age group between 25 and 60 years of age; and
* (5) sign the consent form.

Exclusion Criteria:

* (1) cognitive deficit, evaluated through the Mini Mental State Examination (MMSE);
* (2) illiterate;
* (3) people with metallic implants located on the head, cochlear implants and cardiac pacemaker;
* (4) history of convulsion;
* (5) severe depression, measured by score greater than 36 on Beck Depression Inventory; and
* (6) be pregnant.

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Pain intensity level | Baseline (week 1); Endpoint (week 2 or 3 depending on the arm)
  Changes in pain level, assessed by the Visual Analog Scale, ranges from 0 - 10, with 10 being the highest level of pain.

SECONDARY OUTCOMES:
Quality of life level | Baseline (week 1); Endpoint (week 2 or 3 depending on the arm)
  Changes in quality of life level assessed by Fibromyalgia Impact Questionnaire (FIQ). The FIQ is composed of 19 questions, which measure functional capacity, work status, psychological disturbances, physical and painful symptoms. The greater the impact of the disease, the greater the score found. The FIQ consists of 10 items. The first item contains 10 questions ("a" through "j") related to physical functioning - each issue is evaluated on a four-point Likert scale. In items 2 and 3, the patient is asked to mark the number of days he felt well and the number of days that were unable to work (including housework) because of fibromyalgia-related symptoms. Items 4 to 10 are horizontal lines of 10 cm in length (Visual Analog Scale), in which the patient measures the difficulty for work, pain, fatigue, morning tiredness, stiffness, anxiety and depression.
Health assessment level | Baseline (week 1); Endpoint (week 2 or 3 depending on the arm)
  Changes in health assessed level assessed by Fibromyalgia Health Assessment (HAQ). It has eight categories: clothing and physical presence, wake up, feed, walk, hygiene, reach, footprint and other daily activities. For each of these categories, the patient indicates the degree of difficulty in four possible responses ranging from "no difficulty = 0" to "unable to do it = 3". The score for each category appears in the highest number of any of your items. The final HAQ score is the average of the scores of the eight categories and the higher the final score the worse the test result. Questionaire.
Sleep quality | Baseline (week 1); Endpoint (week 2 or 3 depending on the arm)
  Changes in sleep quality assessed by Pittsburgh Sleep Quality Index.
Cognitive function | Baseline (week 1); Endpoint (week 2 or 3 depending on the arm)
  Changes in the cognitive function assessed by Mini Mental State Examination.
Anxiety level | Baseline (week 1); Endpoint (week 2 or 3 depending on the arm)
  Changes in the anxiety level assessed by Beck Anxiety Inventory
Depression level | Baseline (week 1); Endpoint (week 2 or 3 depending on the arm)
  Changes in the depression level assessed by Beck Depression Inventory
Cortical electrical activity | Baseline (week 1); Endpoint (week 2 or 3 depending on the arm)
  Changes in the cortical electrical activity assessed by electroencephalogram
Resilience | Baseline (week 1); Endpoint (week 2 or 3 depending on the arm)
  Changes in the resilience assessed by Wagnild and Young Resilience Scale. It has 25 items described positively with likert type response ranging from 1 (totally disagree) to 7 (totally agree). Scale scores range from 25 to 175 points, with high values indicating high resilience.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal da Paraiba, João Pessoa, Paraíba, Brazil